CLINICAL TRIAL: NCT07050368
Title: A Phase 1 Translational Study to Assess Brain Activity Using Functional Magnetic Resonance Imaging (fMRI) and to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of MLS101 (Psilocybin) in Healthy Volunteers
Brief Title: A Study Assessing Brain Activity, Safety, Tolerability, and Pharmacokinetics Following Multiple Doses of MLS101 (Psilocybin) in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MycoMedica Life Sciences PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-MLS101-103
Record Dates: First submitted 2025-06-16; First posted 2025-07-03 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MLS101 (Active Comparator)
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — Capsule containing active ingredient, psilocybin
  Arms: MLS101
Drug: Placebo — Capsule with no active ingredients
  Arms: Placebo

SUMMARY:
MLS101 is being developed as a low dose psilocybin, that can be administered to treat neurological and psychiatric conditions.

The purpose of this trial is to investigate brain activity, safety, tolerability, and PK of multiple doses of MLS101 in healthy participants.

DETAILED DESCRIPTION:
In recent years, high-dose psilocybin has gained attention for it potential therapeutic benefit in many psychiatric conditions, however existing clinical data for low psilocybin doses are limited.

The multiple-dose regimen proposed in this study is designed to optimize the pharmacology of MLS101 and elucidate whether it provides a longer period of positive effects, which could be used in future studies in chronic indications such as PMDD, obsessive compulsive disorder and opioid use disorder. Translational functional magnetic resonance imaging (fMRI) imaging will confirm the central nervous system (CNS) activity of priming and repeat low-dose psilocybin, which will serve as a computational evaluation of efficacy and complement the cognitive and perceptual scales and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 55 years old (inclusive) at the time of signing the informed consent form.
* Standard contraception measures are required for this clinical trial.
* Healthy, in the opinion of the Investigator, based on prior (history of) or current (ongoing) medical and psychiatric screening assessments.
* Participants with no clinically significant findings on physical examination, laboratory tests, and cardiac assessment.
* Body mass index (BMI) within the range 18-32 kg/m2, inclusive.
* Normal blood pressure.
* Willing to not operate heavy machinery, including driving a vehicle at least 36 hours post Day 1 dose administration and 24 hours post all other dose administrations.
* Capable of giving signed informed consent which includes the requirements and restrictions as per the approved study protocol

Exclusion Criteria:

* Prior known exposure to psilocybin, LSD, ayahuasca, N, N-Dimethyltryptamine, and related tryptamines, within the past 5 years.
* Prior (history of) or current (ongoing) diagnosis, or first-degree relatives with clinically significant medical or psychiatric condition or disease.
* History of non-hospitalized but medicated Major Depressive Disorder (MDD), Generalized Anxiety Disorder or Panic Disorder ≤ 5 years prior to Screening.
* History of or presence of cardiovascular disease.
* Abnormal and clinically significant ECG.
* Known personal or family history of congenital long QT syndrome or sudden death.
* Current or a history of orthostatic hypotension or postural orthostatic tachycardic syndrome, multiple syncopes, or unresolved/ongoing clinically significant hypotensive episodes or symptoms of fainting, dizziness, or light-headedness.
* History or presence of a neurodegenerative disorder such Alzheimer's disease or Parkinson's disease or other behavioral disturbances resulting from other neurological disorders.
* Use of medications that have CNS effects or affect performance.
* Use of medications with serotonergic activity.
* History or presence of hypersensitivity or idiosyncratic reaction to psilocybin or related compounds or microcrystalline cellulose
* History of substance or alcohol abuse disorder in the last 10 years.
* Participant who, for any reason, is deemed by the Investigator to be inappropriate for this study.
* Contraindications to magnetic resonance imaging (MRI) or fMRI.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI). | Screening to Day 23
  Global functional connectivity
Number and severity of treatment-emergent adverse events (TEAEs) | Screening (Day -90) to end of study visit (Day 44)
  An adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE will be considered treatment-emergent adverse event (TEAE) if the onset date and time is at the time of or after first study drug administration.

SECONDARY OUTCOMES:
Pharmacokinetics of MLS101: area under the plasma concentration-time curve (AUC) | Day 1 to Day 16
  Blood sample collections
Pharmacokinetics of MLS101: maximum observed serum concentration (Cmax) | Day 1 to Day 16
  Blood sample collections
Pharmacokinetics of MLS101: apparent terminal elimination half-life (t½) | Day 1 to Day 16
  Blood sample collections
Pharmacokinetics of MLS101: time corresponding to the occurrence of Cmax (Tmax) | Day 1 to Day 16
  Blood sample collection
Pharmacokinetics of MLS101: apparent total systemic clearance after oral administration (CL/F) | Day 1 to Day 16
  Blood sample collections
Pharmacokinetics of MLS101: apparent volume of distribution during the terminal phase (Vz/F) | Day 1 to Day 16
  Blood sample collections

OTHER OUTCOMES:
Perceptual effects of MLS101 using Mystical Experience Questionnaire (MEQ30) score and change from baseline score. | Day 1 to Day 16
  The MEQ30 consists of 30 questions with each one answered from 0 (none, not at all) to 5 (extreme [more than any other time in my life and stronger than 4]). Full Scale ranges from 0 to 150, with higher scores indicating more psychedelic experience.
Perceptual effects of MLS101 using 5-Dimensional Altered States of Consciousness Rating Scale (5D-ASC) score and change from baseline score. | Day 1 to Day 16
  The 5D-ASC measures altered states of consciousness and contains 94 items using visual analogue scales. Score for each will be calculated from 0 to 100 based on measurement of where the participant has selected on the line. Higher scores mean more altered state of consciousness.
Perceptual effects of MLS101 using the Acute Subjective Effects Scale (ASES) score and change from baseline score. | Day 1 to Day 16
  The Acute Subjective Effects Scale (ASES) is a single question visual analogue scale (VAS) evaluating the present-state intensity of the psychedelic experience on a scale of 0 to 10, where 0 is 'none at all' and 10 is 'most intense'.
Cognitive function: Digit Symbol Substitution Test (DSST) | Day - 1 to Day 16
  The test taker's score is the number of correct symbol-to-number matches they complete within the allotted time. Lower score means worse outcome.
Cognitive function: Trail Making Test A (TMT-A) | Day -1 to Day 16
  The participant draws lines to connect circled numbers in an ascending pattern (i.e., in numerical sequence 1-2-3, etc.) as rapidly as possible. The score is the time it takes the participant to complete the task in seconds. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom